CLINICAL TRIAL: NCT05565846
Title: An Open-Label Study Using NTX-001 to Repair Peripheral Nerve Transection(s)
Brief Title: NTX-001 to Repair Peripheral Nerve Transection(s)
Status: Available | Type: Expanded Access
Sponsor: Neuraptive Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: EA-NTX-22-002
Record Dates: First submitted 2022-07-21; First posted 2022-10-04 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2024-06

CONDITIONS: Peripheral Nerve Transections, Acute or Planned in Upper Extremity and Facial Nerves

STUDY DESIGN:
Expanded Access Types: Intermediate, Treatment

INTERVENTIONS:
Combination Product: NTX-001 — One-time use surgical product of three solutions and a device

SUMMARY:
The proposed use of NTX-001 for transections of upper extremity and facial peripheral nerves, acutely or planned.

DETAILED DESCRIPTION:
For this expanded access program, there is a case-by-case internal review process conducted by Neuraptive after the respective investigator provides a prospective case narrative for enrollment consideration.

Allowed Sunderland Classifications are IV degree (Seddon's Class II) and V degree (Seddon's Class III). If the case is approved, the investigator can move forward.

Patients who are between twelve (12) and eighty (80) years of age and has clinical evidence of a peripheral nerve transection from conditions or interventions that has or may result in motor and/or sensory impairment and require surgical treatment. All peripheral nerve repairs including gap repairs (autografts) will be considered for enrollment.

ELIGIBILITY:
Inclusion:

1. The patient has clinical evidence of a peripheral nerve transection from conditions or interventions that has or may result in motor and/or sensory impairment and requires surgical treatment.

Exclusion:

1. Patients whose nerve repair will occur greater than 48 hours after nerve transection.
2. Patients requiring repair of the intracranial portion of any nerve.
3. Patients requiring a nerve repair involving an allograft or conduit.
4. Patients expected to show signs of spontaneous recovery by 12 months (e.g., Bell's palsy).
5. Patients who, in the judgement of the investigator, are not likely to demonstrate meaningful recovery within a reasonable time frame during follow-up due to significant muscle atrophy or other morbidity.
6. The patient has documented history or clinical signs of any condition where NTX-001 might not prove beneficial (e.g., systemic neuromuscular disease, systemic neurological deficit, or other treatments known to affect the growth and/or physiology of the neural and vascular system).
7. The patient has a known allergy to polyethylene glycol (PEG) or human grade silicone.

Ages: 12 Years to 80 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Orlando Health Orthopedic Institute, Orlando, Florida
  - Harborview Medical Center, Seattle, Washington